CLINICAL TRIAL: NCT06680180
Title: Fibrinolysis Resistance in Infection and Trauma
Acronym: FORTITUDE
Status: Recruiting | Type: Observational
Sponsor: Anders Aneman (Other)
Collaborators: Liverpool Hospital, South Western Sydney Local Health District (Unknown); The Canberra Hospital (Other); Royal North Shore Hospital (Other); Macquarie University, Australia (Other)
Responsible Party: Sponsor-Investigator, Anders Aneman, Conjoint Professor, South West Sydney Local Health District
Organization: South West Sydney Local Health District (Other)
Other Study IDs: 2022/ETH02122
Record Dates: First submitted 2024-10-09; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Sepsis and Septic Shock; Trauma
Keywords: Viscoelastic testing (VET); Sepsis; Trauma; Fibrinolytic Agents; Fibrin Modulating Agents; Tissue Plasminogen Activator; Plasminogen
MeSH Terms: conditions — Sepsis; Shock, Septic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sepsis/Septic shock: According to Sepsis-3 definitions (including SARS CoV-2 as pathogen); expected to remain in ICU and survive beyond the day after tomorrow and for full, active ICU treatment; arterial and secure venous access established or imminent as part of standard care; not on oral anticoagulant/antiplatelet therapy.
  Interventions: Diagnostic Test: Viscoelastometric assessment of fibrinolysis
- Severe Trauma: Admitted via the Emergency Department resuscitation bay requiring trauma team response; deemed at risk of significant blood loss and where transfusion of blood products i considered in the ED during the acute phase of the resuscitation by a senior clinician; expected to remain in ICH and survive beyond the day after tomorrow and for full, active ICU treatment; Not on oral anticoagulant/antiplatelet therapy. A clinical based inclusion approach is the most pragmatic means of patient selection and can be objectively supported by routine blood tests demonstrating poor oxygen supply to the organs. Exclusion criteria: unsurvivable head injury.
  Interventions: Diagnostic Test: Viscoelastometric assessment of fibrinolysis

INTERVENTIONS:
Diagnostic Test: Viscoelastometric assessment of fibrinolysis — Viscoelastometric assessment of whole blood fibrinolysis using supplemental tissue plasminogen activator (tPA) and other agents ex vivo to influence fibrinolysis capacity.

SUMMARY:
Blood coagulation disorders are often seen in critically ill patients e.g. with severe infection or following extensive injury, that can lead to life threatening events as a result of excessive blood clot formation leading to organ failure. This study aims to use Viscoelastic Testing (VET) technology to detect patients at risk of excessive blood blot formation at the bedside, test new blood coagulation drugs, and guide life-saving use of blood modifying treatments.

DETAILED DESCRIPTION:
In healthy individuals blood coagulates (clots) to minimise blood loss then, as part of the process of wound repair, blood clots are broken down in a process called fibrinolysis which involves two key proteins: tissue plasminogen activator (tPA) and plasminogen. In severe infection (sepsis) or following extensive injury (trauma), fibrinolysis abnormalities commonly develop, which include reduced fibrinolysis activity (fibrinolysis resistance) resulting in extensive clot formation and frequently leading to organ failure and death. Currently, the cause of fibrinolysis resistance in sepsis and trauma are unknown and clinical trials to address coagulopathies in sepsis have failed, likely due to inadequate disease phenotyping.

The viscoelastic testing (VET) technology ClotPro® has been used to identify fibrinolysis resistance in 55% of critically ill patients (COVID and non-COVID with acute respiratory failure) and through novel adaptation of the technology, determined that this is likely driven by reduced tPA and/or plasminogen activity. Furthermore, it has been used to detect in real time the impact of a 24 hr tPA infusion on fibrinolysis in a patient. Thus, this preliminary work has demonstrated the feasibility of a personalised treatment approach to fibrinolysis resistance management that can guide life-saving use of fibrinolysis enhancers to overcome resistance in an individualised basis that is likely to increase therapeutic efficacy and safety.

This project aims to scientifically validate the aforementioned preliminary work, increase our knowledge on the mechanisms of reduced fibrinolysis enzyme activity in severe infection and injury, discover potential treatment options, and progress these findings towards translation. The results of this project will drive future clinical trials of repurposed or novel therapies guided by VET to deliver a personalised dose to critically ill patients who demonstrate fibrinolysis resistance, which in conjunction with rapid detection, is anticipated to significantly improve patient outcomes.

ELIGIBILITY:
Sepsis/Septic shock Inclusion Criteria:

* Admission to ICU, needing at least one organ supportand principally for the management of clinically suspected Sepsis or Septic shock according to Spesis-3 criteria (including SARS-COV-2)
* Expected to remain in ICU and survive beyond the day after tomorrow

Sepsis Exclusion Criteria:

* On oral anticoagulant/antiplatelet therapy
* Not for full, active ICU support
* Death is deemed inevitable within 24 hrs

Trauma Inclusion Criteria:

* Trauma is the principal diagnosis on ICU admission
* Expected to remain in ICU and survive beyond the day after tomorrow
* Receiving respiratory support at the time of ICU admission - high-flow nasal prongs, non-invasive or invasive ventilation
* Already received, or considered at risk of needing a blood product transfusion within 24 hrs of injury

Trauma Exclusion Criteria:

* Nursing home resident
* Unsurvivable head injury
* Not for full, active ICU support
* Death is deemed inevitable within 24 hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to an ICU
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
VET testing and analysis | From admission to ICU and at 24 hours, 48 hours, 5 days, 7 days, 10 days, and 15 days post ICU admission
  VET testing in whole blood will determine the kinetics and contribution of:
  i) both plasma and platelets to clot formation following the addition of tissue factor.
  ii) plasma clot formation only by adding tissue factor and platelet inhibitors. iii) tPA-induced fibrinolysis by adding tissue factor and tPA.
  The following test parameters will be used for analytical purposes: clotting time, clot amplitude at 10 min, maximum clot firmness, lysis time, maximum lysis. The platelet contribution to the clot will be calculated by subtracting (ii) from (i). An additional blood sample will be collected at the time of VET analysis for processing and storage for subsequent fibrinolysis protein analysis.
Laboratory evaluation of fibrinolytic profile | From admission to ICU and at 24 hours, 48 hours, 5 days, 7 days, 10 days, and 15 days post ICU admission
  We will evaluate the temporal changes in key fibrinolytic markers (i.e. plasminogen, antiplasmin, PAI-1 activity) and also changes in overall fibrinolytic capacity of patient plasma (i.e. how responsive plasma is to generate plasmin ex vivo) in relation to the VET testing.
  Commercial ELISAs will be used to determine plasminogen, alpha2 antiplasmin levels, PAI-1 and tPA activity; A novel tPA inducible plasmin-antiplasmin test will be used to evaluate plasmin generation; amidolytic assay will be used to determine plasmin activity.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - The Canberra hospital (ICU), Canberra, Australian Capital Territory
  - Liverpool Hospital (ICU), Liverpool, New South Wales
  - Macquarie University Hospital (ICU), Macquarie, New South Wales
  - Royal North Shore Hospital (ICU), St Leonards, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coupland LA, Rabbolini DJ, Schoenecker JG, Crispin PJ, Miller JJ, Ghent T, Medcalf RL, Aneman AE. Point-of-care diagnosis and monitoring of fibrinolysis resistance in the critically ill: results from a feasibility study. Crit Care. 2023 Feb 10;27(1):55. doi: 10.1186/s13054-023-04329-5. PMID 36765421